CLINICAL TRIAL: NCT03050268
Title: Familial Investigations of Childhood Cancer Predisposition
Acronym: SJFAMILY
Status: Recruiting | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SJFAMILY
Record Dates: First submitted 2017-02-08; First posted 2017-02-10 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Acute Leukemia; Adenomatous Polyposis; Adrenocortical Carcinoma; AML; BAP1 Tumor Predisposition Syndrome; Carney Complex; Choroid Plexus Carcinoma; Constitutional Mismatch Repair Deficiency Syndrome; Diamond-Blackfan Anemia; DICER1 Syndrome; Dyskeratosis Congenita; Emberger Syndrome; Familial Acute Myeloid Leukemia; Familial Adenomatous Polyposis; Fanconi Anemia; Familial Cancer; Familial Wilms Tumor; Familial Neuroblastoma; GIST; Hereditary Breast and Ovarian Cancer; Hereditary Paraganglioma-Pheochromocytoma Syndrome; Hodgkin Lymphoma; Juvenile Polyposis; Li-Fraumeni Syndrome; Lynch Syndrome; MDS; Melanoma Syndrome; Multiple Endocrine Neoplasia Type 1; Multiple Endocrine Neoplasia Type 2; Neuroblastoma; Neurofibromatosis Type 1; Neurofibromatosis Type II; Nevoid Basal Cell Carcinoma Syndrome; Non Hodgkin Lymphoma; Noonan Syndrome and Other Rasopathy; Overgrowth Syndromes; Pancreatic Cancer; Peutz-Jeghers Syndrome; Pheochromocytoma/Paraganglioma; PTEN Hamartoma Tumor Syndrome; Retinoblastoma; Rhabdoid Tumor Predisposition Syndrome; Rhabdomyosarcoma; Rothmund-Thomson Syndrome; Tuberous Sclerosis; Von Hippel-Lindau Disease
Keywords: Familial cancer; Genetic predisposition; Heritable disease; Cancer risk; Genome analysis; Genetic modifiers; Next generation sequencing (NGS); Genetic counseling; DNA
MeSH Terms: conditions — Adenomatous Polyposis Coli; Adrenocortical Carcinoma; Carney Complex; Choroid Plexus Carcinoma; Turcot syndrome; Anemia, Diamond-Blackfan; Dyskeratosis Congenita; GATA2 Deficiency; Fanconi Anemia; Hereditary Breast and Ovarian Cancer Syndrome; Hodgkin Disease; Juvenile polyposis syndrome; Li-Fraumeni Syndrome; Colorectal Neoplasms, Hereditary Nonpolyposis; Melanoma; Multiple Endocrine Neoplasia Type 1; Multiple Endocrine Neoplasia Type 2a; Neuroblastoma; Neurofibromatosis 1; Neurofibromatosis 2; Basal Cell Nevus Syndrome; Lymphoma, Non-Hodgkin; Noonan Syndrome; Pancreatic Neoplasms; Peutz-Jeghers Syndrome; Pheochromocytoma; Paraganglioma; Hamartoma Syndrome, Multiple; Retinoblastoma; Rhabdomyosarcoma; Rothmund-Thomson Syndrome; Tuberous Sclerosis; von Hippel-Lindau Disease; Genetic Predisposition to Disease

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, skin or saliva samples and leftover tumor samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
NOTE: This is a research study and is not meant to be a substitute for clinical genetic testing. Families may never receive results from the study or may receive results many years from the time they enroll. If you are interested in clinical testing please consider seeing a local genetic counselor or other genetics professional. If you have already had clinical genetic testing and meet eligibility criteria for this study as shown in the Eligibility Section, you may enroll regardless of the results of your clinical genetic testing.

While it is well recognized that hereditary factors contribute to the development of a subset of human cancers, the cause for many cancers remains unknown. The application of next generation sequencing (NGS) technologies has expanded knowledge in the field of hereditary cancer predisposition. Currently, more than 100 cancer predisposing genes have been identified, and it is now estimated that approximately 10% of all cancer patients have an underlying genetic predisposition.

The purpose of this protocol is to identify novel cancer predisposing genes and/or genetic variants. For this study, the investigators will establish a Data Registry linked to a Repository of biological samples. Health information, blood samples and occasionally leftover tumor samples will be collected from individuals with familial cancer. The investigators will use NGS approaches to find changes in genes that may be important in the development of familial cancer. The information gained from this study may provide new and better ways to diagnose and care for people with hereditary cancer.

PRIMARY OBJECTIVE:

* Establish a registry of families with clustering of cancer in which clinical data are linked to a repository of cryopreserved blood cells, germline DNA, and tumor tissues from the proband and other family members.

SECONDARY OBJECTIVE:

* Identify novel cancer predisposing genes and/or genetic variants in families with clustering of cancer for which the underlying genetic basis is unknown.

DETAILED DESCRIPTION:
During the study, blood samples or other healthy tissue will be obtained from participants, as well as medical and family histories. When possible, leftover tumor samples will also be collected. If participants agree to be re-contacted in the future, they will be asked about once each year to update their health information and family history.

A blood sample will be drawn at St. Jude or at a convenient place of the participant's choice. Saliva collection will be obtained if a blood draw is not possible. For participants who are present at St. Jude, saliva collection will generally be performed only once using a saliva collection kit. However, if the first collection is not sufficient for protocol required studies, then additional saliva samples may need to be collected, for up to a total of 5 occurrences. For non St. Jude participants, or participants who do not wish or cannot come to St. Jude, saliva will be collected locally and shipped back to the St. Jude. A skin sample will be performed as a source of germline DNA from participants who have undergone an allogeneic bone marrow transplant and do not have a source of pre-transplant DNA available. A skin sample will only be obtained one time.

The biological samples will be stored in the St. Jude Biorepository. The DNA of the samples will be studied to determine if there are changes in specific genes that might explain the cancers in the participant or their family members. When available, and if consent is given by the participant, previously collected and stored leftover tumor samples, bone marrow samples or stored DNA may be analyzed.

Genetic variants of interest include: 1) mutations in known genes that may have escaped detection through prior clinical genetic testing; 2) coding mutations predicted to disrupt protein function, particularly in genes and pathways known to be associated with cancer; 3) potential mutations in regulatory regions of the genome, as predicted by epigenetic studies. In some cases, individuals with known predisposing mutations exhibit milder, more severe or atypical phenotypes. Family members who harbor a predisposing mutation but are discordant for a cancer phenotype will be selected for cellular and genetic studies. These will include DNA sequencing and possibly also creation and analysis of induce pluripotent stem cells (iPSC), transcriptome or epigenetic analysis.

All samples will be identified by a code after removal of all personal identifiable information. Samples will remain in the repository for current and future study.

ELIGIBILITY:
NOTE: This is a research study and is not meant to be a substitute for clinical genetic testing. Families may never receive results from the study or may receive results many years from the time they enroll. If you are interested in clinical testing please consider seeing a local genetic counselor or other genetics professional. If you have already had clinical genetic testing and meet eligibility criteria for this study as shown below, you may enroll regardless of the results of your clinical genetic testing.

DEFINITION OF FAMILIAR CANCER FOR THIS PROTOCOL:

In this protocol, the definition of "Familial Cancer" is met if any of the following is present:

* An individual with a history of cancer diagnosed under 26 years of age who has at least one first, second or third degree relative with a history of cancer diagnosed under 51 years of age; OR
* An individual who has been diagnosed with more than one cancer, at least one of which was diagnosed under 26 years of age; OR
* An individual with a clinical or molecular diagnosis of a known cancer predisposition syndrome; OR
* An individual with a congenital cancer diagnosed before 6 months of age; OR
* An individual with a rare pediatric cancer or tumor diagnosed before 26 years of age

º Excluding human papilloma virus-associated cervical cancer and non-melanoma skin cancer occurring in adults.

INCLUSION CRITERIA:

* An individual who meets this protocol's definition of "Familial Cancer," as above.
* Biologic relatives of an individual meeting this protocol's definition of "Familial Cancer," who are either affected or unaffected by cancer.

EXCLUSION CRITERIA:

* An inability or unwillingness of the research participant or his/her legally authorized representative (LAR) to provide written informed consent.
* The participant has received allogeneic bone marrow transplantation and has NO pre-transplant germline (cancer-unaffected) DNA available AND is unwilling to provide a skin sample.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with cancer and their family members who meet the eligibility criteria shown below.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2017-04-06 (Actual); Primary Completion 2037-03-31 (Estimated); Study Completion 2037-03-31 (Estimated)

PRIMARY OUTCOMES:
Identification of novel cancer predisposing genes | Up to 20 years following study activation
  Probands and cancer affected and unaffected relatives from selected families will be sequenced using Whole Genome Sequencing (WGS) or possibly Whole Exome Sequencing (WES) and analyzed to identify new predisposing genetic variants that co-segregate with the tumor phenotype. Data will be analyzed using annotation and filtering strategies to identify potentially deleterious germline mutations that co-segregate with disease.

CONTACTS AND LOCATIONS:
Overall Officials: Kim E. Nichols, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols